CLINICAL TRIAL: NCT02704663
Title: Transumbilical Versus Lateral Transabdominal Removal of Benign Adnexal Masses Via Laparoscopy, a Randomized Trial
Brief Title: Transumbilical Versus Lateral Transabdominal Removal of Benign Adnexal Masses Via Laparoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Päivi Päkarinen, MD PhD, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 98/13/03/03/2014
Record Dates: First submitted 2016-01-18; First posted 2016-03-10 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Postoperative Pain
Keywords: adnexal mass; laparoscopy; removal route; postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transumbilical route (Experimental): Transumbilical removal of benign adnexal masses via laparoscopy.
  Interventions: Procedure: Transumbilical removal of specimen via laparoscopy
- Lateral abdominal route (Active Comparator): Lateral transabdominal removal of benign adnexal masses via laparoscopy.
  Interventions: Procedure: Lateral transabdominal removal of specimen via laparoscopy

INTERVENTIONS:
Procedure: Transumbilical removal of specimen via laparoscopy — Transumbilical removal of a benign adnexal mass from the abdominal cavity in laparoscopy
  Other Names: Transumbilical
  Arms: Transumbilical route
Procedure: Lateral transabdominal removal of specimen via laparoscopy — Lateral transabdominal removal of a benign adnexal mass from the abdominal cavity in laparoscopy
  Other Names: Lateral transabdominal
  Arms: Lateral abdominal route

SUMMARY:
In cases of benign adnexal mass laparoscopic surgery, women were randomized to two groups: transumbilical vs. transabdominal removal. Need for pain medication, postoperative pain and patients´ satisfaction were assessed between the groups, as well as surgeons´ opinions and costs.

DETAILED DESCRIPTION:
Women assigned to laparoscopic surgery for removal of a benign adnexal mass were randomly divided into two groups as regards surgery: a transumbilical (TU) group (n=21) and a transabdominal (TA) group (n=21). General anesthesia and use of local anesthetics were standardized. Visual analog scale (VAS) scores for pain and side effects (nausea/vomiting) and the amount of postoperative analgesic used were recorded for 24 hours. Investigators also investigated the expenses related to endobags and trocars. Further, peri- and postoperative complications were recorded. Investigators inquired about patient satisfaction as well as the surgeons' opinions of the alternative methods available.

ELIGIBILITY:
Inclusion Criteria:

* The criteria for inclusion were scheduled laparoscopy for oophorectomy, salpingo-oophorectomy or cyst enucleation.

Exclusion Criteria:

* The exclusion criteria were contraindications to any of the forms of medication used in the study (oxycodone, ketoprofen, paracetamol),
* language difficulties (inability to understand and speak Finnish or Swedish)
* and suspicion of malignancy.

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2014-11; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
The use of analgesics for postoperative pain | Change in 24 hours after surgery
  The total amount of analgesics used measured by use of Oxycodone (mg)

SECONDARY OUTCOMES:
Complications | The first six months after the surgical intervention
  Frequency of complications. Values are given as n (%) and eventual complications are specified
Nausea | Change in 24 hours after surgery
  Nausea after the procedure: Visual Analog Score (VAS) for nausea, to measure quality of nausea. 10-point VAS score for nausea [(0-10), 0 indicating no nausea and 10 indicating unbearable nausea. at 1, 3, 6, 12 and 24 h (hour) after surgery. (Units on a Scale; 0-10)
Vomiting | Change in 24 hours after surgery
  Vomiting after the procedure: Visual Analog Score (VAS) for vomiting to measure quality of vomiting. 10-point VAS score for vomiting [(0-10), 0 indicating no vomiting and 10 indicating unbearable vomiting] at 1, 3, 6, 12 and 24 h (hour) after surgery. (Units on a Scale; 0-10)
Length of hospital stay in hours | Up to one week
  Length of hospital stay measured from the end of the operation until discharge (hours)
Quality of life | At baseline and 6 months after the surgery
  A questionnaire six months after operation concerning wellbeing outcome after six months (% of respondents in the group)
Cosmetic outcome | At baseline and 6 months after the surgery
  A questionnaire six months after operation concerning cosmetic outcome after six months (% of respondents in the group)
Costs | During the surgery
  Calculating the comparative direct costs of both techniques. The cost of equipment used in the surgical intervention. (euros)
Surgeon perception of both techniques | After one month after the operation
  A questionnaire one month after operation of opinion of surgeons on preferred route of specimen removal (% of respondents in the group)
Length of need of postoperative pain medication | Change in one month after surgery
  A questionnaire of pain medication needed postoperatively. (Days)
Postoperative pain scores | Change in 24 hours after surgery
  Visual Analog Score (VAS) for pain to measure quality of pain. 10-point VAS score for pain [(0-10), 0 indicating no pain and 10 indicating unbearable pain] at 1, 3, 6, 12 and 24 h (hour) after surgery (Units on a Scale; 0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Päivi I Pakarinen, MD PhD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Kätilöopisto Maternity Hospital, Helsinki University hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jokela R, Ahonen J, Tallgren M, Haanpaa M, Korttila K. A randomized controlled trial of perioperative administration of pregabalin for pain after laparoscopic hysterectomy. Pain. 2008 Jan;134(1-2):106-12. doi: 10.1016/j.pain.2007.04.002. Epub 2007 May 15. PMID 17507163
- [Background] Nilsson L, Wodlin NB, Kjolhede P. Risk factors for postoperative complications after fast-track abdominal hysterectomy. Aust N Z J Obstet Gynaecol. 2012 Apr;52(2):113-20. doi: 10.1111/j.1479-828X.2011.01395.x. Epub 2012 Jan 8. PMID 22224504
- [Background] Jokela R, Ahonen J, Tallgren M, Haanpaa M, Korttila K. Premedication with pregabalin 75 or 150 mg with ibuprofen to control pain after day-case gynaecological laparoscopic surgery. Br J Anaesth. 2008 Jun;100(6):834-40. doi: 10.1093/bja/aen098. Epub 2008 Apr 29. PMID 18448418
- [Background] Wodlin NB, Nilsson L. The development of fast-track principles in gynecological surgery. Acta Obstet Gynecol Scand. 2013 Jan;92(1):17-27. doi: 10.1111/j.1600-0412.2012.01525.x. Epub 2012 Nov 1. PMID 22880948
- [Background] Wodlin NB, Nilsson L, Kjolhede P. Health-related quality of life and postoperative recovery in fast-track hysterectomy. Acta Obstet Gynecol Scand. 2011 Apr;90(4):362-8. doi: 10.1111/j.1600-0412.2010.01058.x. Epub 2011 Feb 18. PMID 21306322
- [Background] Alessandri F, Lijoi D, Mistrangelo E, Nicoletti A, Ragni N. Effect of presurgical local infiltration of levobupivacaine in the surgical field on postsurgical wound pain in laparoscopic gynecological surgery. Acta Obstet Gynecol Scand. 2006;85(7):844-9. doi: 10.1080/00016340500494846. PMID 16817084
- [Background] Chou LY, Sheu BC, Chang DY, Huang SC, Chen SY, Hsu WC, Chang WC. Comparison between transumbilical and transabdominal ports for the laparoscopic retrieval of benign adnexal masses: a randomized trial. Eur J Obstet Gynecol Reprod Biol. 2010 Dec;153(2):198-202. doi: 10.1016/j.ejogrb.2010.07.029. Epub 2010 Aug 11. PMID 20705381
- [Background] Ghezzi F, Cromi A, Uccella S, Siesto G, Bergamini V, Bolis P. Transumbilical surgical specimen retrieval: a viable refinement of laparoscopic surgery for pelvic masses. BJOG. 2008 Sep;115(10):1316-20. doi: 10.1111/j.1471-0528.2008.01802.x. PMID 18715419
- [Background] Ghezzi F, Cromi A, Uccella S, Bogani G, Serati M, Bolis P. Transumbilical versus transvaginal retrieval of surgical specimens at laparoscopy: a randomized trial. Am J Obstet Gynecol. 2012 Aug;207(2):112.e1-6. doi: 10.1016/j.ajog.2012.05.016. Epub 2012 May 23. PMID 22704765
- [Background] Akdemir A, Ergenoglu AM, Akman L, Yeniel AO, Sendag F, Oztekin MK. A novel technique for laparoscopic removal of the fallopian tube after ectopic pregnancy via transabdominal or transumbilical port using homemade bag: A randomized trial. J Res Med Sci. 2013 Sep;18(9):777-81. PMID 24381621
- [Background] Kadar N, Reich H, Liu CY, Manko GF, Gimpelson R. Incisional hernias after major laparoscopic gynecologic procedures. Am J Obstet Gynecol. 1993 May;168(5):1493-5. doi: 10.1016/s0002-9378(11)90787-x. PMID 8498433
- [Background] Karthik S, Augustine AJ, Shibumon MM, Pai MV. Analysis of laparoscopic port site complications: A descriptive study. J Minim Access Surg. 2013 Apr;9(2):59-64. doi: 10.4103/0972-9941.110964. PMID 23741110
- [Background] Jansen FW, Kapiteyn K, Trimbos-Kemper T, Hermans J, Trimbos JB. Complications of laparoscopy: a prospective multicentre observational study. Br J Obstet Gynaecol. 1997 May;104(5):595-600. doi: 10.1111/j.1471-0528.1997.tb11539.x. PMID 9166204
- [Background] Marks JL, Ata B, Tulandi T. Systematic review and metaanalysis of intraperitoneal instillation of local anesthetics for reduction of pain after gynecologic laparoscopy. J Minim Invasive Gynecol. 2012 Sep-Oct;19(5):545-53. doi: 10.1016/j.jmig.2012.04.002. Epub 2012 Jul 3. PMID 22763313
- [Background] Yamamoto M, Minikel L, Zaritsky E. Laparoscopic 5-mm trocar site herniation and literature review. JSLS. 2011 Jan-Mar;15(1):122-6. doi: 10.4293/108680811X13022985131697. PMID 21902958